CLINICAL TRIAL: NCT01253616
Title: A Proof-of-Concept Pilot Study Assessing Vagus Nerve Stimulation (VNS) Paired With Tones for Tinnitus
Brief Title: Proof-of-Concept Study Assessing VNS Paired With Tones for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroTransponder Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-T-01
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Severe Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VNS plus tones (Experimental)
  Interventions: Device: vagus nerve stimulation (VNS)

INTERVENTIONS:
Device: vagus nerve stimulation (VNS) — Daily stimulation synchronized with tones at the study assigned dose (amplitude, frequency, on/off cycle and treatment period).

SUMMARY:
This is a proof-of-concept study designed to provide feasibility information on the clinical use of vagus nerve stimulation (VNS) paired with tones for the treatment of severe tinnitus. The study is expected to give preliminary efficacy and safety information.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 65 years of age
* Diagnosed with subjective tinnitus due to hearing loss with at least some tonal quality of the tinnitus.
* Diagnosis of tinnitus for at least one year
* Tinnitus severity of 18 or greater on TRQ cross checked with TQ severity of Grade 3 or worse

Key Exclusion Criteria:

* Acute or intermittent tinnitus
* Severe hearing loss
* History of significant ear disease such as Meniere's disease, ear tumors, or evidence of active middle ear disease.
* Any other implanted device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Audiometric measurements | weekly through one month

SECONDARY OUTCOMES:
tinnitus questionaires | weekly through one month
adverse events | as they occur

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Antwerp, Edegem, Belgium

REFERENCES:
- [Result] De Ridder D, Vanneste S, Engineer ND, Kilgard MP. Safety and efficacy of vagus nerve stimulation paired with tones for the treatment of tinnitus: a case series. Neuromodulation. 2014 Feb;17(2):170-9. doi: 10.1111/ner.12127. Epub 2013 Nov 20. PMID 24255953
- [Result] De Ridder D, Kilgard M, Engineer N, Vanneste S. Placebo-controlled vagus nerve stimulation paired with tones in a patient with refractory tinnitus: a case report. Otol Neurotol. 2015 Apr;36(4):575-80. doi: 10.1097/MAO.0000000000000704. PMID 25689839